CLINICAL TRIAL: NCT03135717
Title: Wasting in Chronic Kidney Disease: Refeeding Techniques and Artificial Nutrition Practices
Brief Title: Wasting in Chronic Kidney Disease
Acronym: PEW
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL14-253
Record Dates: First submitted 2017-04-24; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Chronic Kidney Hospitalized
Keywords: Chronic kidney disease; Enteral nutrition; Oral nutritional supplements; Parenteral nutrition; Refeeding; Wasting
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphagia; Cachexia | interventions — Nutrition Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Nutritional care — * Diagnosis of protein energy wasting : anthropometry, calculation of the nutrient intakes, evaluation of appetite, evaluation of gastrointestinal syndromes, hand grip test and bioimpedancemetry
  * Treatment of protein energy wasting : estimation of nutritional requirements, prescription of oral nutritional supplement or artificial nutrition, physical rehabilitation
  * Multidisciplinary approach (nephrologists, dieticians, physiotherapists, nurses)
  * Evaluation of the nutritional treatment (plasma albumin and prealbumin, weight evolution, muscle strength and body composition)

SUMMARY:
Protein energy wasting is an independent factor associated with morbi-mortality in chronic kidney disease. Wasting is particularly common in chronic diseases of organs such as kidney disease with a major impact at the stage of dialysis. It covers 20 to 70% of patients diagnosed with chronic kidney disease according to the degree of evolution of the disease and the diagnostic method.

Mechanisms of PEW are based mainly on anorexia and metabolic abnormalities caused by kidney disease. Nutritional treatment differs depending on the stage of the kidney disease acute or chronic treated whether or not by dialysis. Nutritional monitoring should be regular, individualized and collaborative to detect a risk of PEW or treat installed PEW. Refeeding techniques should allow all the nutritional needs. Their indications depend on the clinic, biochemical assessment and nutrient intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients with kidney disease
* Patients hospitalized in a university hospital renal ward

Exclusion Criteria:

- Hospitalization less than two weeks

Ages: 44 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Nutritional care evaluated with questionnaire | Since admissions to hospital, up to 4 weeks

SECONDARY OUTCOMES:
body composition | Since admissions to hospital, up to 4 weeks
physical activity | Since admissions to hospital, up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Denis Fouque, Pr, Principal Investigator — Hospices Civils de Lyon